CLINICAL TRIAL: NCT04518436
Title: Diffusion-Weighted Magnetic Resonance Imaging on Surgical Decision-Making in Acute Appendicitis
Brief Title: Diffusion MRI in Appendicitis
Status: Completed | Type: Observational
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Gül Bora Makal, Asist. Prof., Yuksek Ihtisas University
Other Study IDs: observational
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Acute Appendicitis
Keywords: Acute appendicitis; Diffusion weighted magnetic resonance imaging; Diagnostic accuracy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, it was aimed to investigate the effect of diffusion-weighted magnetic resonance imaging on diagnosis and surgical decision in patients with suspected acute appendicitis. Investigators believe that Diffusion-weighted magnetic resonance imaging is a valuable method in the diagnosis of acute appendicitis and in making the decision of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected acute appendicitis and scanned by diffusion weighted magnetic resonance imaging

Exclusion Criteria:

* Patients evaluated by CT
* younger than 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were admitted to the Department of General Surgery and Emergency Medicine with right lower quadrant pain of the abdomen, between January 2015 and May 2019, and scanned by diffusion weighted magnetic resonance imaging
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Diffusion weighted magnetic resonance imaging | preoperative period
  diffusion restriction

CONTACTS AND LOCATIONS:
Overall Officials: Gül BORA MAKAL, Study Director — Asist. Prof.
Locations (1):
- Ankara Medical Park Hastanesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared in a publication when it is possible